CLINICAL TRIAL: NCT03688503
Title: Trial of Magnesium Supplementation and Blood Pressure Reduction Among Adults With Untreated High Blood Pressure
Brief Title: Magnesium Supplementation and Blood Pressure Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Pure Encapsulations (Industry)
Responsible Party: Principal Investigator, Howard D. Sesso, ScD, MPH, Associate Epidemiologist, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018P-001849
Record Dates: First submitted 2018-09-25; First posted 2018-09-28 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Blood Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- magnesium (Active Comparator): magnesium glycinate supplement, 480 mg/day
  Interventions: Dietary Supplement: magnesium glycinate supplement
- placebo (Placebo Comparator): placebo supplement
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: magnesium glycinate supplement — magnesium glycinate (480 mg/day)
  Arms: magnesium
Dietary Supplement: placebo — placebo
  Arms: placebo

SUMMARY:
This double-blind, placebo-controlled randomized clinical trial will test whether a magnesium glycinate supplement (480 mg/day) taken for 12 weeks lowers blood pressure.

DETAILED DESCRIPTION:
This double-blind, placebo-controlled randomized clinical trial will test whether a magnesium glycinate supplement (480 mg/day) taken for 12 weeks lowers blood pressure in 60 adults aged 30-74 who have elevated blood pressure or stage 1 hypertension and are not taking anti-hypertensive medication. Animal studies, epidemiologic studies, and small randomized trials suggest that supplemental Mg may reduce blood pressure, but the evidence is not definitive.

Eligibility to participate in the trial will be determined by a 2-stage screening process -- completion of a pre-screening form online followed by an in-person screening clinic visit. Eligible participants will assigned by chance (like a coin toss) to daily magnesium or to placebo and will receive a supply of study capsules via U.S. mail. Participants will take 4 study capsules per day (2 capsules in the morning and 2 capsules in the evening).

Assessments at the screening visit include seated blood pressure; 24-hour ambulatory blood pressure (monitor will be worn by the participant for 24 hours and then returned via mail); pulse; weight, height, waist and hip circumference measurements; fasting blood and urine collection; and health and diet questionnaires. Participants will return for clinic visits at 6 weeks and at 12 weeks to assess these measures, including 24-hour ambulatory blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of systolic blood pressure 120-139 mmHg or diastolic blood pressure 80-89 mmHg at prescreening
* Measured seated systolic blood pressure 120-149 mmHg or measured seated diastolic blood pressure 80-94 mmHg at screening visit
* Body mass index less than 40 kg/m2
* Total Mg intake from supplements of no more than 100 mg/day
* Willing to maintain current diet and supplement use patterns during the intervention period

Exclusion Criteria:

* History of antihypertensive use
* History of cardiovascular disease (myocardial infarction, stroke, revascularization [coronary artery bypass graft or percutaneous transluminal coronary angioplasty], or angina pectoris)
* History of invasive cancer diagnosed within the last 5 years (non-melanoma skin cancer permitted)
* History of type 1 or 2 diabetes
* History of renal disease
* History of kidney failure
* History of dialysis
* History of pancreatitis
* History of inflammatory bowel disease
* History of hypermagnesemia
* Women who are pregnant, nursing, or intend to become pregnant during the treatment period
* Plan to relocate out of Boston area within the next year
* Unwillingness and/or inability to swallow 4 pills per day
* Inability to provide written informed consent
* Excessive antacid or laxative use within the past 3 months

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Change in seated blood pressure from baseline to 12 weeks | 12 weeks
Change in 24-hour ambulatory blood pressure from baseline to 12 weeks | 12 weeks

SECONDARY OUTCOMES:
Change in plasma renin activity level from baseline to 12 weeks | 12 weeks
Change in angiotensin II level from baseline to 12 weeks | 12 weeks
Change in aldosterone level from baseline to 12 weeks | 12 weeks
Change in creatinine level from baseline to 12 weeks | 12 weeks
Change in high-sensitivity C-reactive protein level from baseline to 12 weeks | 12 weeks
Change in glucose level from baseline to 12 weeks | 12 weeks
Change in insulin level from baseline to 12 weeks | 12 weeks
Change in hemoglobin A1c level from baseline to 12 weeks | 12 weeks
Change in interleukin-6 level from baseline to 12 weeks | 12 weeks
Change in serum magnesium levels from baseline to 12 weeks | 12 weeks
Whether the baseline magnesium status modifies the effect on seated and 24-hour ambulatory BP | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No